CLINICAL TRIAL: NCT01175226
Title: A Phase 2 Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of BTA798 in Asthmatic Adults With Symptomatic Human Rhinovirus Infection
Brief Title: A Phase 2 Study of BTA798 in Asthmatic Adults With Symptomatic Human Rhinovirus Infection
Acronym: RHINO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biota Scientific Management Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Vaxart (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTA798-202
Record Dates: First submitted 2010-08-03; First posted 2010-08-04 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Rhinovirus
Keywords: Human rhinovirus; Aviragen Therapeutics, Inc.; Aviragen Therapeutics; Aviragen
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BTA798 (Experimental)
  Interventions: Drug: BTA798
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BTA798 — BTA798 twice daily
  Arms: BTA798
Drug: Placebo — Placebo twice daily
  Other Names: Glucose
  Arms: Placebo

SUMMARY:
This study aims to evaluate the safety, tolerability and effectiveness of BTA798 on

* shortening the length and reducing the symptoms of human rhinovirus infection (also known as the common cold),
* controlling asthma symptoms, and
* lowering the risk of asthma symptoms worsening in subjects with asthma.

DETAILED DESCRIPTION:
Subjects with a previous diagnosis of asthma will be pre screened within 90 days prior to enrolment. If a subject develops symptoms of human rhinovirus (HRV) infection they will visit the site for assessment. Symptomatic subjects meeting all eligibility criteria will be invited to enroll.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18-70 years
* Diagnosis of asthma consistent with Global Initiative for Asthma (GINA) steps 1 to 3
* Presumptive human rhinovirus infection

Exclusion Criteria:

* Current severe asthma exacerbation
* Severe asthma, GINA steps 4 or higher
* Uncontrolled or clinically significant medical condition, disease or event which could impact subject safety and/or study evaluations and/or compliance to the protocol
* Current smoker, ex-smoker of <1 year, or history of smoking >/=10 pack years.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Lambert, PhD, Study Director — Biota Scientific Management Pty Ltd
Locations (39):
- United States (39):
  - Research Site, Scottsdale, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Fountain Valley, California
  - Research Site, Orange, California
  - Research Site, Waterbury, Connecticut
  - Research Site, Hialeah, Florida
  - Research Site, Bangor, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Papillion, Nebraska
  - Research Site, Albuquerque, New Mexico
  - Research Site, New York, New York
  - Research Site, Newburgh, New York
  - Research Site, North Syracuse, New York
  - Research Site, Rockville Centre, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Lake Oswego, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Upland, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Lincoln, Rhode Island
  - Research Site, Providence, Rhode Island
  - Research Site, San Antonio, Texas
  - Research Site, Waco, Texas
  - Research Site, South Burlington, Vermont
  - Research Site, Richmond, Virginia
  - Research Site, Greenfield, Wisconsin
  - Research Site, Madison, Wisconsin
  - Research Site, West Allis, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BTA798 | Placebo
Started | 155 | 145
Completed | 144 | 140
Not Completed | 11 | 5

BASELINE CHARACTERISTICS:
Population: Safety population - all randomized subjects who received at least 1 dose of investiational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | BTA798 | Placebo | Total
Number analyzed (Participants) | 154 | 145 | 299
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (14.34) | 42.0 (13.69) | 41.3 (14.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 95 | 209
  Male | 40 | 50 | 90
Region of Enrollment [Number; unit: participants]
  United States | 154 | 145 | 299

OUTCOME MEASURES:

1. Primary Outcome: Wisconsin Upper Respiratory Symptom Survey-21 (WURSS-21) Questionnaire
Description: Daily Change in WURSS-21 Severity Score Averaged over Days 2 to 4. The Wisconsin Upper Respiratory Symptom Survey-21 (WURSS-21) Questionnaire is an evaluative illness-specific outcomes instrument designed to assess the severity of cold symptoms and the impact of the common cold (range 0-140), with higher scores indicating more symptoms and functional impairment.
Time Frame: Days 2-4
Population: Intent-to-Treat Infected (ITT-I) Population - all randomized subjects who had a PCR positive result for rhinovirus from nasal swab on Days 1, 3, 5 and 7 with at least 1 post-baseline measurement of efficacy.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | BTA798 | Placebo
Number analyzed (Participants) | 42 | 50
Scores on a scale | -9.12 (1.403) | -5.11 (1.184)
Statistical Analysis 1: Comparison: BTA798 vs Placebo; Test type: Superiority; p = 0.020, ANCOVA

ADVERSE EVENTS:
Description: Adverse events are reported for the Safety Population defined as all randomized subjects who met the eligibility criteria and were randomized.
Arm/Group | BTA798 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/154 | 0/145
Serious Adverse Events (participants affected / at risk) | 0/154 | 0/145
Other Adverse Events (participants affected / at risk) | 22/154 | 18/145
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BTA798 (N=154) | Placebo (N=145)
Headache (Nervous system disorders) | 7 | 6
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 5
Sinusitis (Infections and infestations) | 5 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes